CLINICAL TRIAL: NCT02254161
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Rising Doses of BI 1181181 Given Orally q.d. for 10 Days in Young Healthy Male and Elderly Healthy Male/Female Volunteers (Randomized, Double-blind, Placebo Controlled Within Dose Groups Phase I Study)
Brief Title: Multiple Rising Dose of BI 1181181 Given Orally in Young Healthy Male and Elderly Healthy Male/Female Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1344.2; 2014-002482-30 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Healthy

ARMS (4):
- BI 1181181 healthy young (Experimental): Medium doses as tablets q.d. for 10 days
  Interventions: Drug: BI 1181181 Healthy young
- BI 1181181 healthy elderly (Experimental): Medium doses as tablets q.d. for 10 days
  Interventions: Drug: BI 1181181 healthy elderly
- Matching placebo in healthy young (Placebo Comparator): Matching placebo for 10 days
  Interventions: Drug: Matching placebo
- Matching placebo in healthy elderly (Placebo Comparator): Matching placebo for 10 days
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Matching placebo — Tablet
  Arms: Matching placebo in healthy elderly; Matching placebo in healthy young
Drug: BI 1181181 healthy elderly — Tablet
  Arms: BI 1181181 healthy elderly
Drug: BI 1181181 Healthy young — Tablet
  Arms: BI 1181181 healthy young

SUMMARY:
The primary objective of the current study is to investigate the safety and tolerability of BI 1181181 in healthy young male and elderly male and female volunteers following oral administration of repeated rising doses of BI 1181181, given once daily over 10 days. Secondary objectives are the exploration of the pharmacokinetics (PK) and pharmacodynamics (PD) of BI 1181181.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male or female subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests.
2. Age of 18 to 50 years (incl.) for young healthy volunteers or of 65 to 80 years (incl.) for elderly healthy volunteers.
3. BMI of 18.5 to 29.9 kg/m2 (incl.)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation.

Exclusion criteria:

1. Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
2. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
3. Any evidence of a concomitant disease judged as clinically relevant by the investigator
4. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
5. Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication (except appendectomy)
6. Diseases of the central nervous system (such as epilepsy), other neurological disorders or psychiatric disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
frequency [N (%)] of subjects with drug-related adverse events | days 1 to 24

SECONDARY OUTCOMES:
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval t) after administration of the last dose | 0 to 336 hours
Cmax,ss (maximum measured concentration of the analyte in CSF (if feasible) at steady state over a uniform dosing interval t) after administration of the last dose | 0 to 336 hours
AUCt,1 (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval t after administration of the first dose) | 0 to 336 hours
Cmax (maximum measured concentration of the analyte in plasma) after administration of the first dose | 0 to 336 hours
AUCt,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval t) after the administration of the last dose | 0 to 336 hours
AUCt,ss (area under the concentration-time curve of the analyte in CSF (if feasible) at steady state over a uniform dosing interval t after the administration of the last dose | 0 to 336 hours

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1344.2.1 Boehringer Ingelheim Investigational Site, Berlin, Germany